CLINICAL TRIAL: NCT02439138
Title: Phase II Study of Phosphatidylinositol-3-kinase (PI3K) Inhibitor Idelalisib (GS-1101) in Waldenström Macroglobulinemia
Brief Title: Study of Phosphatidylinositol-3-kinase (PI3K) Inhibitor Idelalisib (GS-1101) in Waldenström Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety issues from trials in CLL
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Jorge J. Castillo, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-040; ISR IN-US-313-1609 (Other Grant/Funding Number: Gilead Sciences, Inc.)
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GS-1101 (Experimental): After the screening procedures confirms eligibility to participate in the research study. Treatment will be administered on an outpatient basis.
  -- Idelalisib (GS-11-01) orally, predetermined dose twice daily per cycle for up to 6 cycles. After this initial 6 month period, for Cycles 7 and beyond, Idelalisib will be administered once a day until disease progression.
  Interventions: Drug: GS-1101

INTERVENTIONS:
Drug: GS-1101 — Oral twice daily for 6 months followed by once daily until disease progression or unacceptable toxicity.
  Other Names: Idealisib; Zydelig; CAL-101

SUMMARY:
This research study is evaluating a drug called idelalisib (formerly known as GS-1101 or CAL-101) as a possible treatment for Waldenstrom's Macroglobulinemia (WM).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug, idelalisib, to learn whether idelalisib works in treating a specific cancer. "Investigational" means that idelalisib is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if idelalisib is effective for treating different types of cancer. Idelalisib has already been approved in the US by the FDA to treat patients with relapsed chronic lymphocytic leukemia, follicular lymphoma and small lymphocytic lymphoma.

Idelalisib is a newly discovered drug that is being developed as an anti-cancer agent. This drug has been used in laboratory experiments and other research studies in B-cell malignancies and information from those other research studies suggests that idelalisib may help to target the tumor cells in B-cell malignancies, including WM. B cells are a type of white blood cell responsible for making antibodies.

In this research study, the investigators are testing the safety and efficacy of idelalisib as a treatment option for relapsed or refractory Waldenstrom's Macroglobulinemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia and meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenstrom's macroglobulinemia (Owen 2003; Kyle 2003).
* Measurable disease, defined as presence of serum immunoglobulin M (IgM) with a minimum IgM level of > 2 times the upper limit of normal of each institution is required.
* Have received at least one prior therapy for WM.
* Age ≥18 years.
* ECOG performance status <2 (see Appendix A.).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count > 1,000/mm3
  * Platelets > 50,000/mm3
  * Hemoglobin > 8 g/dL
  * Total bilirubin ≤1.5 mg/dL or < 2 mg/dL if attributable to hepatic infiltration by neoplastic disease
  * AST (SGOT) and ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine ≤ 2 mg/dL
* Not on any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin.
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study:

  1) while participating in the study; and 2) for at least 28 days after discontinuation from the study. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, uncontrolled intercurrent illness, or psychiatric illness/social condition that would prevent the participant from signing the informed consent form
* Concurrent use of any other anti-cancer agents or treatments or any other study agents
* Prior exposure to idelalisib
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, ECG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the patient; alter the absorption, distribution, metabolism or excretion of Idelalisib; or impair the assessment of study results
* Grade > 2 toxicity (other than alopecia) continuing from prior anti-cancer therapy
* Known central nervous system lymphoma
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening
* New York Heart Association classification III or IV heart failure.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV) infection
* Lactating or pregnant women
* Inability to swallow capsules
* History of non-compliance to medical regimens
* Unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J. Castillo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GS-1101: After the screening procedures confirms eligibility to participate in the research study. Treatment will be administered on an outpatient basis.
  -- Idelalisib (GS-11-01) orally, predetermined dose twice daily per cycle for up to 6 cycles. After this initial 6 month period, for Cycles 7 and beyond, Idelalisib will be administered once a day until disease progression.
  GS-1101
Period: Overall Study
Arm/Group | GS-1101
Started | 5
Completed | 2
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — PI decision to terminate the study | 2

BASELINE CHARACTERISTICS:
Arm/Group | GS-1101
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 66 [57 to 80]
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR measured by decrease in serum IgM level by at least 25% from baseline.
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Population: 4 of 5 participants returned for at least 1 follow-up to assess disease response.
Measure: Number; unit: percentage of participants with response
Arm/Group | GS-1101
Number analyzed (Participants) | 4
percentage of participants with response | 0

2. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Assess the safety and tolerability of idelalisib
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Measure: Number; unit: percentage of participants with AEs
Arm/Group | GS-1101
Number analyzed (Participants) | 5
percentage of participants with AEs | 100

3. Secondary Outcome: Rate of Complete Response (CR)
Description: CR measured by decrease in serum IgM levels to normal range, disappearnace of monoclonal protein by immunofixation, no evidence of bone marrow involvement, and resolution of any extramedullary disease by CT scan.
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Measure: Number; unit: percentage of participants with CR
Arm/Group | GS-1101
Number analyzed (Participants) | 4
percentage of participants with CR | 0

4. Secondary Outcome: Rate of Very Good Partial Response (VGPR)
Description: VGPR measured by decrease in serum IgM levels of at least 90% from baseline.
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Measure: Number; unit: percentage of participants with VGPR
Arm/Group | GS-1101
Number analyzed (Participants) | 4
percentage of participants with VGPR | 0

5. Secondary Outcome: Rate of Partial Response (PR)
Description: PR measured by decrease in serum IgM levels of between 25% and 50% from baseline.
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Measure: Number; unit: percentage of participants with PR
Arm/Group | GS-1101
Number analyzed (Participants) | 4
percentage of participants with PR | 0

6. Secondary Outcome: Rate of Minimal Response
Description: Minimal response measured by decrease in serum IgM levels of between 25% and 50%.
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Measure: Number; unit: percentage of participants with MR
Arm/Group | GS-1101
Number analyzed (Participants) | 4
percentage of participants with MR | 0

7. Secondary Outcome: Rate of Stable Disease
Description: Stable disease measured by serum IgM levels <25% reduced from baseline.
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Measure: Number; unit: percentage of participants with SD
Arm/Group | GS-1101
Number analyzed (Participants) | 4
percentage of participants with SD | 100

8. Secondary Outcome: Rate of Progressive Disease
Description: Progressive disease measured by an 25% increase in serum IgM level with an absolute increase of at least 500mg/dL from the lowest attained IgM on therapy.
Time Frame: Participants were followed for the duration of therapy, a median of one cycle, for up to 3 cycles.
Measure: Number; unit: percentage of participants with PD
Arm/Group | GS-1101
Number analyzed (Participants) | 5
percentage of participants with PD | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of screening until 30 days post treatment discontinuation, up to 16 weeks (median 4 weeks).
Arm/Group | GS-1101
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GS-1101 (N=5)
INR elevation (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
ALT elevation (Investigations) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GS-1101 (N=5)
Headache (Nervous system disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Thrush (Investigations) | 1 (1)
Sweats (General disorders) | 1 (1)
Shaking chills (General disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Painful gums (General disorders) | 1 (1)
AST elevation (Investigations) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mouth sores (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to safety concerns from the previously untreated CLL experience. All participants who remained on study at that time were permanently removed from protocol therapy. The median time on protocol therapy was 1 cycle

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No